CLINICAL TRIAL: NCT06558851
Title: The Effect of Systematic Endurance Training in Treatment of Women With Lipedema - The LipidEx Study
Brief Title: The Effect of Systematic Endurance Training in Treatment of Women With Lipedema
Acronym: LipidEx
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St.Olavs Hospital, Trondheim University Hospital, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 795836
Record Dates: First submitted 2024-07-10; First posted 2024-08-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The exercise intervention group perform three sessions of HIIT per week for 12 weeks. HIIT involves 4 times 4-minutes intervals at 85-95% of maximal heart rate (HRmax) with 3-minutes active breaks (~60% HRmax) between the intervals. Two HIIT sessions are supervised at the NextMove core facility, and performed on treadmills or spinning bikes, while the last session of HIIT is unsupervised. In this unsupervised session, HIIT in a pool will be recommended based on the potential benefits gained from compression. The criteria for adequate compliance to the exercise intervention program will be set to ≥80%.
  Interventions: Behavioral: High intensity endurance training
- Control (No Intervention): In the control period, the participants will live as normal.

INTERVENTIONS:
Behavioral: High intensity endurance training — 12 weeks of high intensity endurance training three times a week. Two of the weekly sessions are supervised.
  Arms: Exercise

SUMMARY:
Lipedema is a chronic adipose tissue disorder that primarily affects women. The etiology remains unclear and involves abnormal buildup of fat mainly in the lower limbs. It causes physical and psychological morbidity, often with significant impact of daily life. Effective treatment options are still limited, primary involving conservative measures such as compression therapy. Regular endurance training is known to have positive effects on pain management in other disorders, as well as beneficial effects on obesity management. Thus, LipidEx aims to explore the potential of high-intensity interval training (HIIT) as a novel therapeutic option for women with lipedema. We will now perform a cross-over randomized controlled trial (RCT) exploring the effects of 12 weeks of HIIT compared to a control period of usual care. Primary outcomes include changes in pain, and secondary outcomes include changes in adipose tissue mass and quality of life. Exploratory outcomes include changes in inflammatory markers, metabolites, and lipoprotein subfractions in blood and adipose tissue.

DETAILED DESCRIPTION:
Design This study will follow the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) reporting guidelines.

Study design and participants We will conduct a crossover randomized controlled trial (RCT) involving 58 women diagnosed with lipedema. To be eligible for participation, women must be between 18 and 65 years old and have a confirmed diagnosis of lipedema. Exclusion criteria include ongoing eating disorders and orthopedic limitations that prevent exercise training. Eligible participants will be randomized (1:1) using block randomization in eForsk to either the exercise intervention group or the control group. The exercise intervention group will undergo 12 weeks of high-intensity interval training (HIIT), tailored to each participant's fitness level and the severity of their lipedema. The control group will continue their usual lifestyle during this period. Following the 12-week intervention, there will be a 12-week wash-out period during which all participants will resume their normal activities. After the wash-out period, participants will switch groups, allowing all included participants to receive the exercise intervention and potentially experience the benefits of HIIT. In total, the study duration for each participant will be 9 months.

Recruitment Patients will be recruited in Trøndelag, Norway, primarily through The Clinic of Rehabilitation at St. Olavs Hospital and the social media channels of the Norwegian Lymphedema and Lipedema Foundation (NLLF). Additionally, posters will be displayed at general practitioner offices and various physiotherapy clinics in the Trondheim area. Eligible patients will receive comprehensive information about the study and will be given at least one week to consider their participation.

Exercise intervention Exercise testing and training will be conducted at state-of-the-art exercise training facility at the Norwegian University of Science and Technology (NTNU), the NextMove Core facility, supported by highly experienced staff. The exercise intervention group perform three sessions of HIIT per week for 12 weeks. HIIT involves 4 times 4-minutes intervals at 85-95% of maximal heart rate (HRmax) with 3-minutes active breaks (~60% HRmax) between the intervals. Two HIIT sessions are supervised at the NextMove core facility, and performed on treadmills or spinning bikes, while the last session of HIIT is unsupervised. In this unsupervised session, HIIT in a pool will be recommended based on the potential benefits gained from compression. The criteria for adequate compliance to the exercise intervention program will be set to ≥80%. With standardized templated from the NextMove core facility, the participants are required to write a diary of their physical activity during the entire study period, including the exercise intervention period, the wash-out period, and the control period.

Data collection During the first study visit, participants will be randomized into groups and receive comprehensive information about the study and all included procedures. Data collection will occur primarily on four separate test days: before and after both the exercise intervention period and the control period. On these test days, anthropometric and physiological measurements will be taken, questionnaires will be completed, and fasting blood samples and tissue biopsies will be collected.

General information, including details on lipedema (type and stage, and time of diagnosis), comorbidities, sleep patterns, and the use of medications, supplements, and clinical aids (e.g., compression aids and their frequency of use), will also be gathered.

Each test day will last approximately three hours. During this time, fasting blood samples and anthropometric measurements will be taken first, followed by a light meal, completion of questionnaires, and performance of physiological measurements. Additionally, participants who consent to adipose tissue biopsies will have two samples collected: one within five days before the first exercise session and one within five days after the final exercise session.

Pain registration Pain will be registered before and after both the intervention period and the control period using the RAND-36 health survey (Pain Dimension) (primary endpoint). RAND-36 (also known as SF-36) includes two questions designed to measure the intensity of pain and the extent to which pain interferes with normal work (both outside the home and housework). One of the questions assess the intensity of pain experienced over the past four weeks with six response options from "none" to "very severe". The second question evaluates the degree to which pain has interfered with daily activities and work with five response options from "not at all" to "extremely". In addition, pain will be registered before and after both the intervention period and the control period using the questionnaire Brief Pain Inventory (BPI). This questionnaire includes four questions that assess the severity of pain right now and at its worst, least, and average. Each question gives a possible answer of 0 to 10, were 0 means no pain and 10 is the worst pain you can imagine. The four BPI questions contribute with the same weight, and they are combined to a final pain severity score with a range from 0 to 40. The results from RAND-36 and BPI will be evaluated separately. While both tools assess pain, the BPI provides a deeper and more detailed assessment of pain characteristics and functional impact compared to the broader, more generalized assessment provided by the RAND-36 pain dimension. However, the questionnaires focus on different timeframes, as RAND-36 assesses pain over a retrospective period of the past 4 weeks whereas BPI assess pain over the past 24 hours or at the present moment (current pain intensity). Potentially, RAND-36 can be more useful for assessing chronic pain, and BPI for assessing more chronic pain, however, the best tool for assessing pain in lipedema is currently unknown.

Anthropometric measurements Body composition, including weight (kg), body mass index (kg/m2), muscle mass (kg), adipose tissue mass (%), basal metabolic rate (kcal), and mineral status (kg), will be measured non-invasively using the bioimpedance instrument InBody 770 (Biospace CO, Ltd, Seul, Korea). The instrument provides both total adipocyte mass and adipose tissue mass in the lower limbs (secondary endpoints). The heigh (m) will be measured without shoes. The circumference (cm) of the waist, hip, right calf, and right thigh will be measured with standard procedures at NextMove, and the waist-to-hip ratio (cm/cm) will be calculated. A measuring board will be used to ensure similar site for pre- and post-measurement of the right calf and thigh.

Quality of life The RAND-36 questionnaire will be used to detect potential changes in health-related quality of life during the study period (secondary endpoint). This questionnaire includes 36 questions covering eight health domains, including vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each domain is scored on a scale from 0 to 100, where the scaled scores are weighted sums of all questions within each of the eight domains. A higher score indicates better health and well-being.

Physiological measurements Blood pressure will be measured in a sitting position after minimum five minutes rest in a quiet room with a handheld sphygmomanometer (Tycos, 5098-02CB, USA) by trained personnel. At the pre- and post-tests, the blood pressure will be measured at the same time-point of the day for each participant. The first reading will be discarded and the mean of the next three consecutive readings will be used. Additional readings will be required if the coefficient of variation is above 15%.

Maximal oxygen uptake (VO2max) will be measured using ergospirometry (Metalyzer ll, Cortex Biophysik GmBH, Leipzig, German) supervised by qualified personnel. To demonstrate cardiometabolic effects from the HIIT intervention, VO2max will be measured during uphill treadmill walking or running. A 10-minute warm-up (~60% of HRmax) will be performed before increasing the workload (speed or incline) every minute until exhaustion. The criteria for reaching VO2max is a levelling off oxygen uptake (VO2) despite increased workload, and a respiratory exchange ratio of ≥1.05. HR will be measured continuously during the test with Polar belt and watch (Polar, Polar Electro, Kempele, Finland), and the data will be used to determine HRmax.

Blood samples and adipose tissue biopsies Four fasting venous blood samples will be drawn by qualified personnel and by standard in-hospital procedures at St.Olavs Hospital. Directly after collection, one 3mL EDTA-tube and one 3mL Li-heparin-tube will be sent to routine biochemical analyses at St. Olavs hospital for such as glucose, HbA1C, triglycerides, HDL-cholesterol, total cholesterol, serum ferritin and hs-CRP. The two remaining tubes (serum and EDTA) will be centrifuged, aliquoted, and stored in the LipidEx biobank at -80°C for explorative analyses.

Two adipose tissue biopsies will be collected by experienced personnel from the Research outpatient clinic at St.Olavs Hospital before and after the exercise intervention. The collected adipose biopsies will be used to advance our physiological understanding of exercise-induced effects on adipose tissue in lipedema patients. To ensure patient comfort during the procedure, local anesthesia will be administered at the site of biopsy to minimize pain and discomfort associated with the needle insertion. The proposed methodology will adhere to rigorous sterilization protocols, including the use of sterile equipment, gloves, and disinfection procedures. A fine needle is used to avoid the need for extensive incisions and to reduce patient discomfort and recovery time. One biopsy will be snap-frozen in liquid nitrogen and stored at -80°C for later explorative analyses. Another biopsy will be placed in histology cassettes and fixed in 4% formaldehyde in 0.1 M phosphate buffer for 24 hours. The samples will be dehydrated, embedded in paraffin, sectioned, and stained at the general lab at the Institute for Circulation and Medical Imaging, NTNU in later explorative analyses.

ELIGIBILITY:
Inclusion Criteria:

Confirmed lipedema diagnosis

Exclusion Criteria:

Ongoing eating disorders and/or orthopedic limitations for exercise training

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain levels | Through study completion, an average of 8 weeks
  Pain will be registered before and after both the intervention period and the control period using the RAND-36 health survey (Pain Dimension) (primary endpoint). RAND-36 (also known as SF-36) includes two questions designed to measure the intensity of pain and the extent to which pain interferes with normal work (both outside the home and housework). One of the questions assess the intensity of pain experienced over the past four weeks with six response options from "none" to "very severe". The second question evaluates the degree to which pain has interfered with daily activities and work with five response options from "not at all" to "extremely". I

SECONDARY OUTCOMES:
Adipose tissue mass | Through study completion, an average of 8 weeks
  Total adipose tissue mass and adipose tissue mass in the lower limbs measured by bioimpedance.
Health-related quality of life | Through study completion, an average of 8 weeks
  Measured by RAND-36

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Rognmo, Study Director — Norwegian University of Science and Technology
Locations (1):
- Institute for Circulation and Medical Imaging, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes